CLINICAL TRIAL: NCT06815926
Title: Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Efficacy of a Probiotic Product in Weight Control
Brief Title: Clinical Trial to Evaluate the Effect of a Probiotic Product on Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioithas SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Probi.Obes
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Overweight, Obesity Grade I
Keywords: probiotics; overweight; obesity; food supplement; gut microbiota
MeSH Terms: conditions — Overweight; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PROBIOTIC (Experimental)
  Interventions: Dietary Supplement: Probiotic
- PLACEBO (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Food supplement based on probiotics in capsule format. Dose: 1 capsule/day.
  The active capsules contain probiotic strains at ≥1×10^9 cfu/dose and excipient.
  Arms: PROBIOTIC
Dietary Supplement: Placebo — Food supplement in capsule format. Dose: 1 capsule/day.
  The placebo capsules contain only excipient (probiotics are not included).
  Arms: PLACEBO

SUMMARY:
The study of the intestinal microbiota and its relationship with health and disease, as well as the use of probiotics as effective alternative treatments to improve people's well-being is a field of growing research in recent years.

Overweight and obesity are increasingly common due to the current lifestyle, but this is not incompatible with the growing interest of the population in taking care of themselves, both physically and psychologically, and, in general, the interest in food supplements, including those based on probiotics, is increasingly common.

The objective of the clinical trial is to evaluate the effectiveness of a food supplement based on probiotics to reduce body weight in 104 volunteers with overweight and type I obesity (BMI 25 - 34.9 kg/m2).

This randomized, double-blind and placebo-controlled clinical trial has a 12-week intervention period, during which subjects have to take a daily dose of the product (probiotic or placebo).

In this trial, anthropometric clinical data, the effect of the intervention on blood parameters and the composition of the intestinal microbiota will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years.
* Body Mass Index (BMI) between 25.0 and 34.9 (overweight or obesity type I).
* Commitment to maintaining a lifestyle, including diet and sports habits, constant throughout the study.
* Signing of informed consent.

Exclusion Criteria:

* Subjects with diabetes (type I or II), hypothyroidism or other diseases that may promote weight gain.
* Presence of other serious pathologies, including cancer or autoimmune diseases, or any other that, at the medical discretion of the investigator, may influence the results of the study.
* Subjects who have participated in a weight loss program or who have substantially modified their lifestyle habits (diet, physical exercise) during the previous 3 months.
* Treatment with antibiotics in the previous 4 weeks.
* Consumption of products or drugs intended for weight loss or satiety control, or that may influence weight in the previous 4 weeks.
* Consumption of products containing probiotics in the previous 2 months.
* Contraindication to taking the product under investigation, or allergy or intolerance to any of its ingredients.
* In the case of women: pregnancy or breastfeeding, or plans to become pregnant during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-07-03 (Actual); Study Completion 2025-07-03 (Actual)

PRIMARY OUTCOMES:
Changes in body weight between baseline and 6- and 12-weeks | Baseline, 6-week and 12-week
Changes in body mass index (BMI) baseline and 6- and 12-weeks | Baseline, 6-week and 12-week

SECONDARY OUTCOMES:
Changes in waist/hip circumference ratio between baseline and 6- and 12-weeks | Baseline, 6-week and 12-week
Changes in body composition between baseline and 12-weeks | Baseline and 12-week
  Body composition is assessed by DEXA (Dual-Energy X-ray Absorptiometry). Lean mass and fat mass of the different body regions will be measured as grams (g) and percentage (%).
Changes in blood pressure between baseline and 6- and 12-weeks | Baseline, 6-week and 12-week
Changes in gut microbiota composition between baseline and 12-weeks | Baseline and 12-week
  Alpha diversity, beta diversity and bacterial taxonomic composition of the gut microbiota will be assessed by sequencing the 16S rRNA gene of stool samples.
Changes in the score of gastrointestinal symptoms questionnaire between baseline and 6- and 12-weeks | Baseline, 6-week and 12-week
  Questionnaire with 15 questions related to gastrointestinal discomfort during the last month.
  Each question is valued according to: None = 1; Insignificant = 2; Mild = 3; Moderate = 4; Quite strong = 5; Strong = 6; and Very strong = 7.
  The total score is calculated by adding the number of answers answered for the different degrees of discomfort (1-7), and is between 15 and 105 points. The higher the score, the worse the indication of gastrointestinal symptoms.
Changes in the score of International Physical Activity Questionnaire (IPAQ) between baseline and 12-weeks | Baseline and 12-week
  International Physical Activity Questionnaire (IPAQ) measures the time spent being physically active during the past 7 days.
  The type of activity is divided into: vigorous activity, moderate activity, walking, and no activity (sitting).
  Weekly activity is recorded in Mets (Metabolic Equivalent of Task or Metabolic Rate Units) per minute and week. The reference Mets values are:
  * Walking: 3.3 Mets.
  * Moderate physical activity: 4 Mets.
  * Intense physical activity: 8 Mets. To obtain the total number of Mets, the reference Mets values are multiplied by the time in minutes of performing each type of activity in a day and by the number of days per week that it is performed.
  Depending on the number of Mets, physical activity is categorized as high, moderate, or low.
Changes in the MEDiterranean LIFEstyle index (MEDLIFE) questionnaire between baseline and 12-weeks | Baseline and 12-week
  The MEDiterranean LIFEstyle index (MEDLIFE) consists of 28 questions categorized into three blocks: 1. Consumption of Mediterranean foods (15 questions); 2. Mediterranean dietary habits (7 questions); and 3. Physical activity, rest, social habits and coexistence (6 questions).
  Each question is scored with 0 or 1 point depending on whether or not it meets the established criteria, so the total score is between 0 and 28 points (the higher the score, the greater the adherence to the Mediterranean lifestyle).
Changes in the score of the Simplified Nutritional Appetite Questionnaire (SNAQ) between baseline and 12-weeks | Baseline and 12-week
  Simplified Nutritional Appetite Questionnaire (SNAQ)
  The questionnaire consists of 4 questions.
  The results are scored on the following numerical scale: a 1, b 2, c 3, d 4, e 5. The sum of the scores for the individual items constitutes the SNAQ score. The total score ranges from 5 to 20 points.
Changes in blood count between baseline and 12-weeks | Baseline and 12-week
  Values of complete blood count.
Changes in glucose levels between baseline and 12-weeks | Baseline and 12-week
  Blood glucose values.
Changes in insulin levels between baseline and 12-weeks | Baseline and 12-week
  Blood insulin values.
Changes in glycosylated hemoglobin (HbA1c) levels between baseline and 12-weeks | Baseline and 12-week
  Blood glycosylated hemoglobin (HbA1c) values.
Changes in LDL and HDL, and total cholesterol levels between baseline and 12-weeks | Baseline and 12-week
  Blood LDL and HDL, and total cholesterol values.
Changes in triglycerides levels between baseline and 12-weeks | Baseline and 12-week
  Blood triglycerides values.
Changes in creatinine and urea levels between baseline and 12-weeks | Baseline and 12-week
  Blood creatinine and urea values.
Changes in AST/GOT and ALT/GPT levels between baseline and 12-weeks | Baseline and 12-week
  Blood AST/GOT and ALT/GPT values.
Changes in C-reactive protein levels between baseline and 12-weeks | Baseline and 12-week
  Blood C-reactive protein values.
Changes in leptin levels between baseline and 12-weeks | Baseline and 12-week
  Blood leptin values.

OTHER OUTCOMES:
Adverse events (AEs) | 6-week and 12-week
  AEs reported by participants, whether or not related to the intake of the investigational products, including required pharmacological treatments if applicable.
Adherence rate to the investigational product | 6-week and 12-week
  Adherence is assessed through leftover capsules and days between visits.

CONTACTS AND LOCATIONS:
Locations (1):
- MiBioPath Research Group (UCAM), Murcia, Spain